CLINICAL TRIAL: NCT07045012
Title: The Relationship Between Osteoporosis and Sarcopenia Parameters in Postmenopausal Women Under 60: A Cross-Sectional Study
Brief Title: The Relationship Between Osteoporosis and Sarcopenia Parameters in Postmenopausal Women Under 60
Status: Not yet recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, Principle Investigator, Beylikduzu State Hospital
Other Study IDs: Beylikdüzüstateh20
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This cross-sectional study will include postmenopausal women under the age of 60 who visited the Physical Medicine and Rehabilitation outpatient clinic at Beylikdüzü State Hospital between June 25 and July 25, 2025. Participants must have undergone a bone mineral density (BMD) assessment within the past six months using Dual X-ray Absorptiometry (DXA). Both osteoporotic and non-osteoporotic patients will be enrolled. Sociodemographic data such as age, height, weight, and BMI will be recorded. Femoral neck and L1-L4 T-scores and BMD values will be obtained from existing DXA results. Information on osteoporosis treatment, presence of fecal incontinence, constipation, and medication use will be collected. In the second phase, sarcopenia will be assessed according to EWGSOP2 criteria using bioelectrical impedance analysis for skeletal muscle mass, handgrip strength, and the five-time sit-to-stand test. Differences between the osteoporotic and non-osteoporotic groups will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Women under 60 years of age who are postmenopausal.
* Patients with or without a diagnosis of osteoporosis:

Osteoporosis group: T-score ≤ -2.5 in femoral neck or L1-L4 region. Control group: T-score ≥ -1.0 in femoral neck and L1-L4 region.

-Patients who provide written informed consent to participate in the study.

Exclusion Criteria:

* Refusal to participate in the study.
* Presence of neuromuscular diseases that could cause muscle loss.
* History of infection, recent surgery, or trauma.
* Presence of psychiatric disorders.
* Cognitive impairment that could interfere with test performance or data reliability.
* Use of medications that could affect study outcomes (e.g., corticosteroids, muscle relaxants, or medications influencing bone/muscle metabolism).

Ages: 50 Years to 59 Years | Sex: Female
Age Groups: Adult
Study Population: Postmenopausal women under 60 years
Sampling Method: Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2025-07-25 (Estimated); Study Completion 2025-07-25 (Estimated)

PRIMARY OUTCOMES:
Skeletal Muscle Mass | 0 day
  Measured by bioelectrical impedance analysis (BIA), this assesses the amount of muscle tissue in the body. Low skeletal muscle mass indicates sarcopenia.
Handgrip Strength | 0 day
  This is a simple test to measure muscle strength. Reduced handgrip strength is a sign of sarcopenia.
5 times chair stand test | 0 day
  The Five Times Sit-to-Stand Test is a simple and widely used functional assessment tool to evaluate lower extremity muscle strength, balance, and mobility.